CLINICAL TRIAL: NCT01155323
Title: Proclear 1 Day Lens vs 1-Day Acuvue Moist Daily Disposable Contact Lens Crossover Study
Brief Title: Two Week Cross-Over Study Comparing Two Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Johnson & Johnson K.K. Medical Company (Industry); Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0926; DISP-523 (Other: Visioncare Research Ltd)
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Results first posted 2011-10-04 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- etafilcon A/omafilcon A (Active Comparator): etafilcon A contact lenses will be worn during the first week and omafilcon A contact lenses will be worn during the second. Lenses were replaced daily
  Interventions: Device: etafilcon A; Device: omafilcon A
- omafilcon A/etafilcon A (Active Comparator): omafilcon A contact lenses will be worn during the first week and etafilcon A contact lenses will be worn during the second. Lenses were replaced daily.
  Interventions: Device: etafilcon A; Device: omafilcon A

INTERVENTIONS:
Device: etafilcon A — 1-day soft contact lens
Device: omafilcon A — 1-day soft contact lens

SUMMARY:
This study seeks to evaluate and compare the clinical performance of two daily disposable soft contact lenses, Proclear 1 Day and 1-Day Acuvue Moist.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and no more than 39 years of age
* Existing soft contact lens wearers
* Willing to signed a written Informed Consent.
* Own a mobile phone and are willing to receive and reply to Short Message Service (SMS) messages during the day.
* Have a contact lens spherical distance requirement between -1.00 diopters (D) and -6.00 diopters (D) in both eyes.
* Have an Astigmatism of 1.00D or less in both eyes.
* Require a visual correction in both eyes.
* Be correctable to a visual acuity of 6/9 (20/30) or better in each eye.
* Have normal eyes with no evidence of abnormality or disease that would preclude lens wear.

Exclusion Criteria:

* Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, tarsal abnormalities, bulbar infection, or any other abnormality of the cornea that would contraindicate contact lens wear.
* Clinically significant corneal staining (Grade 3 in more than one region).
* Keratoconus or other corneal irregularity.
* Abnormal lachrymal secretions.
* Extended wear of contact lenses last 3 months.
* Polymethyl methacrylate (PMMA) or rigid gas-permeable (RGP) lens wear in the previous 8 weeks.
* Refractive surgery.
* Eye injury/surgery within 8 weeks immediately prior to enrollment for this study.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Require concurrent ocular medication
* Any systemic illness which would contraindicate lens wear or the medical treatment of which would affect vision or successful lens wear.
* Any infectious disease (e.g., hepatitis, tuberculosis) or any immunosuppressive disease (e.g., HIV).
* Diabetes.
* Pregnant, lactating or planning a pregnancy at the time of enrollment.
* Participation in any concurrent clinical trial or in last 30 days.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2010-06-01 (Actual); Study Completion 2010-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny Sim, Diploma in Optometry, Principal Investigator — Singapore Polytechnic
Locations (1):
- Singapore Plytechnic, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- Etafilcon A/Omafilcon A: etafilcon A contact lenses will be worn first and omafilcon A contact lenses will be worn second.
- Omafilcon A/Etafilcon A: omafilcon A contact lenses will be worn first and etafilcon A contact lenses will be worn second.
Period: First Intervention
Arm/Group | Etafilcon A/Omafilcon A | Omafilcon A/Etafilcon A
Started | 60 | 58
Completed | 59 | 57
Not Completed | 1 | 1
Not completed — exclusion criteria | 1 | 1
Period: Second Intervention
Arm/Group | Etafilcon A/Omafilcon A | Omafilcon A/Etafilcon A
Started | 59 | 57
Completed | 58 | 56
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total Number of Participants: This represents all subjects that completed the study minus one additional subject excluded due the discovery after study completion that the subject conflicted with exclusion criteria.
Arm/Group | Total Number of Participants
Number analyzed (Participants) | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 33
Region of Enrollment [Number; unit: participants]
  Singapore | 113

OUTCOME MEASURES:

1. Primary Outcome: Subjective Rating of Comfort
Description: This outcome is a weighted combined score calculated from individual comfort-related questions asked on a 1-5 scale: 1 = most negative response to 5 = most positive response.
Time Frame: after 1 week of lens wear
Population: The analysis population represents subjects that completed the study per protocol.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Etafilcon A; Omafilcon A: soft contact lens replaced daily, worn for one week.
Arm/Group | Etafilcon A | Omafilcon A
Number analyzed (Participants) | 113 | 113
Units on a scale | 3.33 (0.09) | 3.32 (0.09)
Statistical Analysis 1: Comparison: Etafilcon A vs Omafilcon A; The alternative hypothesis was that etafilcon A would be superior to omafilcon A for comfort; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.21 to 0.23], Standard Error of Mean 0.11 — Mean difference is calculated as etafilcon A minus omafilcon A

2. Primary Outcome: Vision Quality
Description: This outcome is a weighted combined score calculated from individual vision-related questions asked on a 1-5 scale: 1 = most negative response to 5 = most positive response.
Time Frame: after 1 week of lens wear
Population: The analysis population represents subjects that completed the study per protocol.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Etafilcon A | Omafilcon A
Number analyzed (Participants) | 113 | 113
Units on a scale | 3.53 (0.08) | 3.50 (0.08)
Statistical Analysis 1: Comparison: Etafilcon A vs Omafilcon A; The alternative hypothesis was that etafilcon A would be non-inferior to omafilcon A for vision; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -0.50; Mixed Models Analysis; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.19 to 0.25], Standard Error of Mean 0.11 — The mean difference is calculated as etafilcon A minus omafilcon A

3. Primary Outcome: Subjective Rating of Handling
Description: This outcome is a weighted combined score calculated from individual lens handling-related questions asked on a 1-5 scale: 1 = most negative response to 5 = most positive response.
Time Frame: after 1 week of lens wear
Population: The analysis population represents subjects that completed the study per protocol.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Etafilcon A | Omafilcon A
Number analyzed (Participants) | 113 | 113
Units on a scale | 3.48 (0.09) | 3.48 (0.09)
Statistical Analysis 1: Comparison: Etafilcon A vs Omafilcon A; The alternative hypothesis was that etafilcon A would be non-inferior to omafilcon A for lens handling; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -0.50; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.22 to 0.22], Standard Error of Mean 0.11 — The mean difference is calculated as etafilcon A minus omafilcon A

4. Primary Outcome: Corneal Staining
Description: Investigator assessment of the corneal staining. Staining is an indication of dryness on areas on the cornea. Here it is measured over 5 regions of the cornea: central, temporal, nasal, inferior, and superior. The staining is graded using the National Eye Institute (NEI)0-3 scale: grade 0 = normal, grade 1 = mild, grade 2 = moderate, grade 3 = severe.
Time Frame: after 1 week of lens wear
Population: The analysis population represents subjects that completed the study per protocol.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Etafilcon A | Omafilcon A
Number analyzed (Participants) | 113 | 113
Units on a scale | 0.07 (0.01) | 0.09 (0.01)
Statistical Analysis 1: Comparison: Etafilcon A vs Omafilcon A; The alternative hypothesis was that etafilcon A would be equivalent to omafilcon A for corneal staining; Test type: Non-Inferiority or Equivalence — Margin = +/-0.50; Mixed Models Analysis; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.03 to 0.01], Standard Error of Mean 0.01 — The mean difference is calculated as etafilcon A minus omafilcon A

5. Primary Outcome: Subjective Rating of Quality Perceptions
Description: This outcome is a weighted combined score calculated from individual quality perception-related questions asked on a 1-5 scale: 1 = most negative response to 5 = most positive response.
Time Frame: after 1 week of lens wear
Population: The analysis population represents subjects that completed the study per protocol.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Etafilcon A | Omafilcon A
Number analyzed (Participants) | 113 | 113
Units on a scale | 3.51 (0.08) | 3.44 (0.08)
Statistical Analysis 1: Comparison: Etafilcon A vs Omafilcon A; The alternative hypothesis was that etafilcon A would be non-inferior to omafilcon A for quality perceptions; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -0.50; Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.15 to 0.29], Standard Error of Mean 0.11 — The mean difference is calculated as etafilcon A minus omafilcon A

6. Primary Outcome: Limbal Hyperemia
Description: This outcome is assessed by the investigator during biomicroscopy examination using the following 0-4 scale: 0 = none, 1 = trace, 2 = mild, 3= moderate, 4 = severe.
Time Frame: after 1 week of wear
Population: The analysis population represents subjects that completed the study per protocol.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Etafilcon A | Omafilcon A
Number analyzed (Participants) | 113 | 113
Units on a scale | 0.51 (0.02) | 0.48 (0.02)
Statistical Analysis 1: Comparison: Etafilcon A vs Omafilcon A; The alternative hypothesis was that etafilcon A would be equivalent to omafilcon A from limbal hyperemia; Test type: Non-Inferiority or Equivalence — Margin = +/- 0.50; Mixed Models Analysis; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.01 to 0.06], Standard Error of Mean 0.02 — The mean difference is calculated as etafilcon A minus omafilcon A

ADVERSE EVENTS:
Arm/Group | Etafilcon A | Omafilcon A
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/116
Other Adverse Events (participants affected / at risk) | 0/116 | 0/116

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may not be published or publicly presented without prior written approval of the sponsor. If the investigator wishes to publish or present any study findings, investigator shall contact sponsor to discuss publication plan.